CLINICAL TRIAL: NCT05442944
Title: Analysis of the Impact of Uncomplicated Physiotherapeutic Procedures on the Correlation of Static and Dynamic Balance and the Speed of Reaction in the Elderly - a Randomized Observational Study
Brief Title: Dynamic and Static Balance and the Speed of Reaction in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, Principal Investigator, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9/KRN/2011
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2022-06

CONDITIONS: Spondyloarthritis
Keywords: elderly,; physiotherapy,; static balance,; dynamic balance,; reaction speed,; risk of falls
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A study group with physiotherapeutic intervention. (Experimental): The study group - 30 people - participated in the three-week physiotherapy program.
  Interventions: Procedure: Physiotherapeutic procedures
- A Control group without physiotherapeutic intervention (No Intervention): The control group - 30 people - did not participate in the program.

INTERVENTIONS:
Procedure: Physiotherapeutic procedures — As part of the rehabilitation program, the patients performed two exercises in the Universal Therapeutic Rehabilitation Room (UTRR) system. The patient's task was to perform simultaneous abduction and adduction of the upper and lower limbs. The duration of the procedure was 10 minutes, the patient performed the exercises at a comfortable pace. In the second exercise - the patient's task was to alternately bend and straighten the opposite lower and upper limbs. The duration of the exercise was 10 minutes. The combined duration of both procedures used was 20 minutes. In addition, each patient underwent three physical therapy treatments. The procedures were carried out 5 days a week (Monday to Friday) for three weeks.
  Arms: A study group with physiotherapeutic intervention.

SUMMARY:
The balance of the body in the elderly is disturbed for various reasons and relatively often.

The aim of our research was to analyze the effect of five simple physiotherapeutic procedures on the reaction speed as well as static and dynamic balance in the elderly.

60 people (women and men diagnosed with degenerative changes of the spine, chronic period of the disease) aged 65-95 years were analyzed. Patients were randomly assigned to the study group (30 people - participating in the three-week physiotherapy program) and the control group (30 people - not participating in the program). The test consisted in checking the state of static (postural stability) and dynamic (risk of falls) balance on the Biodex SD dynamic platform and the assessment of speed in the Timed Up-and-Go (TUG) test. The results of our research showed that five simple physiotherapy treatments can significantly improve the reaction speed and the dynamic and static balance in the sagittal plane in the elderly.

DETAILED DESCRIPTION:
The balance of the human body is the result of a properly developed musculoskeletal system, an efficiently functioning nervous system and labyrinth, organs of deep feeling, and the organ of vision. The speed of reaction is an important factor in maintaining the body's balance and reduces the risk of falls, not only in the elderly.

The aim of the study is to analyze the influence of uncomplicated physiotherapeutic procedures on the reaction speed as well as static and dynamic balance in the elderly.

60 people (degenerative changes of the spine) in the chronic period of the disease were analyzed. Age of respondents: 65-95 years, women and men. Patients were randomly assigned to the study group (30 people - participating in the three-week physiotherapy program) and the control group (30 people - not participating in the program). The test consisted in checking the state of static (postural stability) and dynamic (risk of falls) balance on the Biodex SD dynamic platform. Additionally, each patient participated in the Timed Up-and-Go (TUG) test. In the study group, most of the studied variables, analyzed before and after rehabilitation, differed significantly (frontal plane inclinations p = 0.024; QuadsL p = 0.002; TUG p = 0.022). Significant differences were also noted between the groups after the end of the therapy (QuadsL 1 p = 0.015; PostL p = 0.011). Moreover, the correlation between TUG and anterior and lateral (p = 0.032) was confirmed. Conclusions: The use of simple physiotherapeutic procedures significantly improves the reaction speed as well as dynamic and static balance in the sagittal plane in the elderly. Improvement in sagittal static stability and deterioration in the coronal plane contribute to a reduction in TUG time.

ELIGIBILITY:
Inclusion Criteria:

* 1) age over 65, 2) generalized degenerative disease, 3) osteoarthritis of the lumbar spine, 4) possibility of walking at least 6 meters without orthopedic support, 5) ability to stand up and sit on a chair independently.

Exclusion Criteria:

* 1) other than the required disease entity, 2) neurological diseases, labyrinth diseases, vascular imbalances, 3) use of psychotropic drugs, 4) cognitive disorders, 5) people who do not meet the requirements of the equipment used for measurements (weight over 136 kg, height under 130 cm, height over 178 cm), 6) high, low blood pressure, dizziness, malaise.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2012-03-14 (Actual)

PRIMARY OUTCOMES:
Postural stability - static balance on Biodex SD dynamic platform. | Before therapy
  Postural stability was investigated by forward deflections in the sagittal plane.
Postural stability - static balance on Biodex SD dynamic platform. | Before therapy
  Postural stability was investigated by backward deflections in the sagittal plane.
Postural stability - static balance on Biodex SD dynamic platform. | Before therapy
  Postural stability was investigated sideways, in the frontal plane.
Postural stability - static balance on Biodex SD dynamic platform. | Before therapy
  Postural stability was investigated by inward deflections in the frontal plane.
Risk of falls - dynamic balance on Biodex SD dynamic platform. | Before therapy
  The evaluation of the dynamic equilibrium was carried out by measuring the mean deviations of the center of gravity of the subject (overall) on an unstable substrate, the lability of which varied with time, from a more stable state to unstable ground. The Biodex SD platform has a twelve-point instability scale, where level 12 corresponds to a rigid and stable setting and level 1 to a hypermobility setting. For the purposes of the study, levels from 8 to 4 were used.
Speed of reaction as measured by the functional Timed Up and Go (TUG) test. | Before therapy
  The task of the subject during the test was, on the command "start" given by the examiner, to perform the following activities as soon as possible: get up from the chair, walk three meters straight, go around the cone, return the same way to the place, and sit on the chair again. The investigator measured the time of all performed motor tasks from giving the command and starting them until returning to the chair.
Postural stability - static balance on Biodex SD dynamic platform. | Before therapy
  Percent of the time spent by the center of body mass in individual quadrants of the platform.

SECONDARY OUTCOMES:
Postural stability - static balance on Biodex SD dynamic platform. | After 3 weeks of therapy
  Postural stability was investigated by forward deflections in the sagittal plane.
Postural stability- static balance on Biodex SD dynamic platform | 3 weeks after therapy
  Postural stability was investigated by backward deflection in the sagittal plane
Postural stability - static balance on Biodex SD dynamic platform. | 3 weeks after therapy
  Postural stability was investigated sideways, in the frontal plane.
Postural stability - static balance on Biodex SD dynamic platform. | 3 weeks after therapy
  Postural stability was investigated by inward deflections in the frontal plane.
Risk of falls - dynamic balance on Biodex SD dynamic platform. | 3 weeks after therapy
  The evaluation of the dynamic equilibrium was carried out by measuring the mean deviations of the center of gravity of the subject (overall) on an unstable substrate, the lability of which varied with time, from a more stable state to an unstable ground. The Biodex SD platform has a twelve-point instability scale, where level 12 corresponds to a rigid and stable setting and level 1 to a hypermobility setting. For the purposes of the study, levels from 8 to 4 were used.
Speed of reaction as measured by the functional Timed Up and Go (TUG) test. | 3 weeks after therapy
  The task of the subject during the test was, on the command "start" given by the examiner, to perform the following activities as soon as possible: get up from the chair, walk three meters straight, go around the cone, return the same way to the place, and sit on the chair again. The investigator measured the time of all performed motor tasks from giving the command and starting them until returning to the chair.
Postural stability - static balance on Biodex SD dynamic platform. | 3 weeks after therapy
  Percent of the time spent by the center of body mass in individual quadrants of the platform.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olczak, PhD, Principal Investigator — Rehabilitation Clinic, Military Institute of Medicine